CLINICAL TRIAL: NCT00805610
Title: The Use of Human Hepatocyte Transplantation as a Life Support Bridge in Terminal Liver Failure.
Brief Title: Hepatocyte Transplantation in Liver Failure
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Investigator taking position at another university-0 enrolled under this protocol.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCU IRB 124
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Liver Failure
Keywords: Liver Failure; Hepatocyte Transplantation; Liver Transplantation
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hepatocyte Transplantation (Experimental): Hepatocyte Transplantation through single donor will be transplanted into the liver via intraportal or intrasplenic routes.
  Interventions: Biological: Hepatocyte Transplantation

INTERVENTIONS:
Biological: Hepatocyte Transplantation — Briefly, prepared hepatocytes from a single donor will be transplanted into the liver via intraportal or intrasplenic routes.

SUMMARY:
The investigators research will examine the safety and efficacy of hepatocyte transplantation in the patient with acute liver failure without history of chronic disease. The investigators will study the effectiveness in providing a bridge of support for patient survival until whole organ transplantation is possible. This support may also be a bridge to recovery; by allowing the native liver to recover so that orthotopic liver transplant is not necessary.

The investigators will also study the safety and efficacy of hepatocyte transplantation in the patient with chronic liver disease. Underlying etiologies of chronic disease may arise from cirrhosis, fibrosis or inherited metabolic disorders. The investigators will examine cell transplantation in end-stage patients not eligible for whole organ transplant. These patients may benefit with an amelioration of symptoms that will allow other therapeutic treatments.

The investigators study will also examine the ability of transplanted hepatocytes to treat inherited metabolic diseases (ex., Crigler-Najjar Disease, Familial Hypercholesterolemia, Urea Cycle Disorders). Cell transplant may also act as a 'bridge' to whole organ transplant or improve function, permitting easier disease control through traditional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are specific to the classification of liver disease, i.e., fulminant or non-fulminant or metabolic disease

Exclusion Criteria:

* Any systemic infection
* Unstable coronary artery disease
* HIV infection
* Preformed antibodies to class antigens that are present on all available donor samples (Only cells from an ABO-compatible donor with no HLA Class I antigen to which the recipient has preformed antibodies will be selected for transplant.)
* Hepatopulmonary disease (Room air Pa02 ≤ 60 mmHg)
* Testing positive for Hepatitis B Surface Antigen (HBsAg), Hepatitis Be antigen (HBeAg) or Hepatitis B Virus by DNA and unable to receive or pay for Hepatitis B treatment.
* Any current or anticipated contraindication for the use of tacrolimus and cyclosporine, methylprednisolone or prednisone.
* Female patients who are breast feeding
* Any medical condition that, in the opinion of the investigator, makes the patient unsuitable for participation in this trial.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The functional capability of transplanted hepatocytes to assume function in the native liver. | Outcome measurements will be assessed weekly through week two post transplant, then monthly through month 12, then every six months.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Fisher, M.D., Principal Investigator — Virginia Commonwealth University Health System
Locations (1):
- Virginia Commonwealth University Health System, Richmond, Virginia, United States